CLINICAL TRIAL: NCT03582111
Title: Ultrasound Diagnosis of Cleft Lip and Palate - FENCHU
Brief Title: Ultrasound Diagnosis of Cleft Lip and Palate
Acronym: FENCHU
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0284
Record Dates: First submitted 2018-06-27; First posted 2018-07-10 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-06

CONDITIONS: Cleft Lip and Palate
Keywords: Ultrasound; Pregnancy; Diagnosis
MeSH Terms: conditions — Cleft Lip; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women who have a foetus with a cleft lip/palate: Pregnant women who have a foetus with a cleft lip/palate
  Interventions: Other: Study of medical records

INTERVENTIONS:
Other: Study of medical records — Study of medical records

SUMMARY:
Cleft lips and palate are one of the most frequent congenital malformation. From 2005 to 2009, a French study, conducted by Dr Bäumler et al. evaluated the accuracy of prenatal ultrasound in the diagnosis of cleft palate when cleft lip is present.

The aim of this study is to continue this study from 2009 till 2016. The hypothesis is that the diagnosis rate is constant since 2005.

ELIGIBILITY:
Inclusion criteria:

* Age over 18
* Prenatal ultrasound diagnosis of cleft palate/lip.
* Viable pregnancy or Intrauterine fetal demise or medical termination of pregnancy

Exclusion criteria:

- Diagnosis not confirmed at birth and ultrasound picture not interpretable

Ages: 18 Years to 46 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Fœtus with cleft lip diagnosed at mid-trimester ultrasound screening in Montpellier hospital (Arnaud de Villeneuve) between February 2009 and December 2016.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2009-02 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Compare the prenatal and postnatal diagnosis of cleft lip and palate | At birth
  Compare the prenatal and postnatal diagnosis of cleft lip and palate

SECONDARY OUTCOMES:
Study the cleft palate diagnosis when cleft lip is present | At birth
  Study the cleft palate diagnosis when cleft lip is present

CONTACTS AND LOCATIONS:
Overall Officials: Cyrielle LEFEBVRE, Midwife, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC